CLINICAL TRIAL: NCT00706810
Title: Combination of Hydroxyurea and Verapamil for Refractory Meningiomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI25089
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Cancer; Brain Cancer; Meningioma
Keywords: Cancer; Brain cancer; Meningioma
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Meningioma | interventions — Hydroxyurea; Verapamil

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental)
  Interventions: Drug: Hydroxyurea; Drug: Verapamil

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea inhibits DNA synthesis by inhibition of ribonucleotide diphosphate reductase and is a well-known drug used for the treatment of a number of tumor types including head and neck tumors and chronic myelogenous leukemia. It has also been used as an adjuvant for antiretroviral treatment for patients with HIV and as a treatment for polycythemia vera, essential thrombocythemia and sickle cell disease.
Drug: Verapamil — Verapamil is another commonly used medication. It is used for the treatment of angina, hypertension, supraventricular arrhythmias, and migraine prophylaxis. Dosing with standard verapamil is 80-120 mg pox three times a day but the sustained release form can be given 120-480mg once or twice each day.

SUMMARY:
Meningiomas account for 20% of primary adult brain tumors, occurring at an annual incidence of 6 per 100,000 (Louis, Scheithauer et al. 2000). Complete surgical resection is the treatment of choice but may not possible when the tumor invades critical structures (e.g., skull base, sagittal sinus) (Mirimanoff, Dosoretz et al. 1985; al-Rodhan and Laws 1990; Al-Rodhan and Laws 1991; Newman 1994; De Monte 1995; Levine, Buchanan et al. 1999; Barnett, Suh et al. 2000; Ragel and Jensen 2003). Up to 20% of meningiomas exhibit a more aggressive phenotype that does not respond to standard therapies (Kyritsis 1996). Adjuvant therapies are critical for patients with this subset of meningiomas. Radiation therapy and stereotactic radiosurgery are good adjuvant therapies but are limited by radiation neurotoxicity, tumor size constraints, and injury to adjacent vascular structures or cranial nerves (Goldsmith, Wara et al. 1994; Barnett, Suh et al. 2000; Goldsmith and Larson 2000). Standard chemotherapeutic treatments have been disappointing (Kyritsis 1996). Even drugs like temozolomide that have shown efficacy against malignant brain tumors have failed to inhibit the growth of refractory meningiomas in a phase II study (Chamberlain, Tsao-Wei et al. 2004).

DETAILED DESCRIPTION:
The investigators have demonstrated previously that the calcium channel antagonists (CCAs) verapamil, nifedipine, and diltiazem can block in vitro and in vivo meningioma growth at clinically relevant doses (Jensen, Lee et al. 1995; Jensen, Petr et al. 2000; Jensen and Wurster 2001). However, only modest growth inhibition was exhibited in the tumors in these studies with CCAs alone. Many authors have shown augmented growth inhibition by adding CCAs to traditional chemotherapies in other tumor types (Tsuruo, Iida et al. 1981; Tsuruo, Iida et al. 1983; Helson 1984; Robinson, Clutterbuck et al. 1985; Ince, Appleton et al. 1986; Merry, Fetherston et al. 1986; Cano-Gauci and Riordan 1987). For instance, the combination of verapamil and 1,3-bis (2-chloroethyl)-1-nitrosourea (BCNU) is better than BCNU alone in inhibiting the growth of human gliomas in vitro and in vivo (Bowles, Pantazis et al. 1990). Calcium antagonists seem to exert the majority of their anti-tumor effects by inhibiting calcium dependent secondary messenger systems (Metcalfe, 1986 #74; Jensen, 2000 #15). Furthermore, the investigators have more recently demonstrated that the addition of a verapamil or diltiazem with HU enhances the growth inhibition seen with these drugs in vitro and in vivo.

Hydroxyurea inhibits DNA synthesis by inhibition of ribonucleotide diphosphate reductase and is a well-known drug used for the treatment of a number of tumor types including head and neck tumors and chronic myelogenous leukemia. It has also been used as an adjuvant for antiretroviral treatment for patients with HIV and as a treatment for polycythemia vera, essential thrombocythemia and sickle cell disease.

Hydroxyurea is well absorbed after oral administration with the peak serum concentration achieved in two hours. The drug is excreted primarily in the urine, either as urea or as the unchanged compound. The drug is supplied as 500 mg capsules in a white crystalline powder. It is stored at room temperature. Dosing is usually in the range of 20 mg/kg/day with adjustments necessary for patients with renal insufficiency. In the current study population patients would be usually treated with 500mg twice a day. It is contraindicated in patients with myelosuppression or severe anemia.

Verapamil is another commonly used medication. It is used for the treatment of angina, hypertension, supraventricular arrhythmias, and migraine prophylaxis. Dosing with standard verapamil is 80-120 mg pox three times a day but the sustained release form can be given 120-480mg once or twice each day. It is contraindicated in patients with left ventricular dysfunction, congestive hart failure, hypotension (systolic <90bpm) 2nd or 3rd degree atrioventricular block (except in patients with a functioning artificial pacemakers), or sick sinus syndrome and atrial flutter or atrial fibrillation and an accessory bypass tract (Wolff-Parkinson-White Syndrome, Lown-Ganong-Levine Syndrome). Serious adverse reactions associated with Verapamil use are congestive heart failure, hypotension, bradycardia, 2nd or 3rd degree AC block, angina, myocardial infarction, syncope and GI obstruction.

STUDY PROCEDURES:

Screening and pretreatment assessments: Written informed consent is obtained before study-specific screening evaluations are performed. After receiving a subject's agreement to participate in the study and verifying that the subject meets eligibility criteria, the following will be performed: Medical and surgical history, prior cancer therapy (including prior chemotherapy and radiation therapy), complete physical examination, orthostatic vital signs, blood pressure, heart rate, temperature, weight, height, Karnofsky performance status (See appendix), neurological evaluation, current medications, and drug allergies. The following laboratory evaluations will be obtained: complete blood count (including differential, hemoglobin, and platelet count), serum chemistries (BUN, creatine, sodium, potassium, bicarbonate, chloride, calcium, glucose, LDH, total protein, total bilirubin, ALT, AST, alkaline phosphatase, albumin), serum pregnancy test (for woman of childbearing age, for all other women - documentation in the medical history will confirm that the subject is not of childbearing potential). All subjects will undergo an ECG test at screening. Patients with incomplete bundle branch or first degree AV conductions problems that don't exclude them from the study will be monitored with serial monthly ECG exams or more frequently if symptoms occur. All subjects will undergo an MRI of the brain (or CT with contrast if unable to do MRI) with and without Gadolinium contrast to assess tumor measurements within three to four weeks prior to beginning treatment. Patients will also undergo Positron Emission Tomography (PET) with metabolic FDG (radiopharmaceutical fluorodeoxyglucose) markers to assess tumor activity. Baseline FDG/PET scans will be given to all enrolled patients at screening and every 6 months, thereafter.

Assessments during treatment phase: Patients receive oral hydroxyurea twice daily for 2 years in the absence of disease progression or unacceptable toxicity. Responders may continue beyond the 2 years of protocol treatment at the discretion of the physician. If the therapy is stopped for any reason, therapy may be reinstituted if the discontinuance does not exceed 4 consecutive weeks. The dose is 20 mg/kg/day divided in twice daily doses. The calculated dose will be rounded up or down to the nearest multiple of 500 mg. Patients will typically receive either 1,000 mg/day or 1,500 mg/day. If the dose is 1,500 mg/day, it should be divided as 500 mg po every morning and 1,000 mg po. at bedtime. Verapamil sustained release tablets will begin at a dose of 120 mg each day for two weeks, then 240 mg each day for two weeks, then 360 mg each day for two weeks, then 240 mg twice a day. If the baseline SBP is <110 mmHg then the initial Verapamil sustained release dose will be 60 mg (1/2 of a 120 mg tablet) each day for two weeks. Patients will have blood pressure and heart rate measurements done weekly for the first month and them monthly thereafter. Other clinical and laboratory evaluations will be performed at 1 month intervals and include: limited physical examination, orthostatic vital signs, blood pressure, heart rate, temperature, Karnofsky performance status, neurologic evaluation, serum chemistries (BUN, creatine, sodium, potassium, bicarbonate, chloride, calcium, glucose, LDH, total protein, total bilirubin, ALT, AST, alkaline phosphatase, albumin). Concomitant medications and adverse events will also be collected. Complete blood counts (including differential, hemoglobin, and platelet count), will be done weekly throughout the study until counts stabilize for two months, and then labs will be done every two weeks thereafter to closely monitor the side-effect of myelosuppression.

Patients with incomplete bundle branch or first degree AV conduction abnormalities that don't exclude them from the study will be monitored with monthly ECG exams or more frequently if symptoms occur. Subjects will undergo MRI with gadolinium (or CT with contrast if unable to do MRI) every three months after beginning treatment. Measurements will be made of the image slice with the largest cross sectional area. Two orthogonal measures will be made to determine maximal AP and lateral dimensions. PET imaging will be done at baseline and every 6 months and proliferative and metabolic activity will be compared to baseline images. Tumor location and tumor size will be obtained by CT/MRI. Treatment response and clinical progression can frequently be difficult to measure directly. Serial neurological exams, CT/MRI and PET scans may provide a guide to the actual course of response and progression. Deterioration in neurological status and tumor regrowth on CT/MRI and PET must be sustained over time to declare clinical progression. The time interval until progression will be measured from the day of last CT/MRI before treatment and every 3-4 months until deterioration is documented. The patient should consistently be followed with the same diagnostic imaging study and formal evaluation of radiological tumor progression and tumor response will be done post study

Patients will be treated for up to two years on the study. Progression of disease will be defined as a greater than 25% increase of largest cross sectional area by two orthogonal measurements. Patients will be discontinued for illness that prevents further treatment including unacceptable toxicity (Grade 3 or 4 that fails to resolve with dose medication per protocol) of study drugs.

ELIGIBILITY:
1. Must be age > 18 years
2. Patient able to provide written informed consent
3. Histologically confirmed meningioma of any WHO grade (written pathology report from surgery required)
4. Radiographic demonstration of at least 25% increase in tumor cross sectional area measured on CT/MRI within last 6 months
5. Patients refusing or for which there is no further surgical or radiation therapy options
6. WBC at least 2,500/mm3
7. Platelet count of at least 100,000/mm3
8. Hemoglobin > 8.0 g/dL
9. Renal insufficiency (glomerular filtration rate (GFR) < 60 as estimated by the Cockcroft-Gault equation) are ineligible
10. Hepatic disease (ALT, AST, bilirubin, or alkaline phosphatase > 3 times upper limit of normal) or known cirrhosis are ineligible
11. Clinically significant cardiovascular disease specifically those patients with the following conditions are ineligible:

    * congestive heart failure
    * known bundle branch or AV conduction problems
    * 2nd or 3rd degree atrioventricular block (except in patients with artificial pacemaker),
    * sick sinus syndrome
    * atrial flutter or atrial fibrillation with an accessory bypass tract (Wolff-Parkinson-White Syndrome, Lown-Ganong-Levine Syndrome),
    * history of myocardial infarction in the past 6 months
    * currently taking beta-blockers, digoxin, or neuromuscular blocking agents
    * Bradycardia (resting heart rate < 60 beats per minute)
12. Hypotension (resting blood pressure < 90 systolic)
13. Altered neuromuscular transmission (Duchenne Muscular Dystrophy, myasthenia gravis)
14. Karnofsky performance score 50-100%
15. Life expectancy more than 6 months
16. Pregnant or nursing females are ineligible. Fertile patients must use an effective contraception
17. Received prior investigational agents in the past 6 months are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Jensen, MD, Ph.D., Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Karsy M, Hoang N, Barth T, Burt L, Dunson W, Gillespie DL, Jensen RL. Combined Hydroxyurea and Verapamil in the Clinical Treatment of Refractory Meningioma: Human and Orthotopic Xenograft Studies. World Neurosurg. 2016 Feb;86:210-9. doi: 10.1016/j.wneu.2015.09.060. Epub 2015 Sep 30. PMID 26428319

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Groups
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 50 [25 to 76]
Sex/Gender, Customized [Number; unit: participants]
  Female | 6
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Serious Adverse Events Including But Not Limited to Hospitalizations, Deaths Related to Treatment, or Other Incapacitating Conditions.
Description: Adverse Events assessed in accordance with CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 3.0.
Time Frame: two years
Measure: Number; unit: participants
Arm/Group | All Groups
Number analyzed (Participants) | 7
participants | 0

2. Secondary Outcome: Median Progression-free Survival Rates of the Treatment Population.
Description: Response and progression will be evaluated in this study using measurements from the MRI/CT scans. Measurements will be made of the image slice with the largest cross sectional area. Two orthogonal measures will be made to determine maximal AP and lateral dimensions. Progression of disease will be defined as a greater than 25% increase of largest cross sectional area by two orthogonal measurements, taking as reference the smallest sum recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 31 months
Measure: Median (Full Range); unit: months
Arm/Group | All Participants
Number analyzed (Participants) | 7
months | 8.0 [5 to 31]

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=7)
abdominal pain (Gastrointestinal disorders) | 1
anemia (Blood and lymphatic system disorders) | 5
back pain (Musculoskeletal and connective tissue disorders) | 1
constipation (Gastrointestinal disorders) | 3
decreased eye acuity (Eye disorders) | 1
dizziness (Nervous system disorders) | 2
ear infection (Infections and infestations) | 1
edema (Vascular disorders) | 1
fatigue (General disorders) | 2
headache (Nervous system disorders) | 1
heart palpatations (Cardiac disorders) | 1
hypocalcemia (Metabolism and nutrition disorders) | 1
hyponatremia (Metabolism and nutrition disorders) | 1
leukopenia (Blood and lymphatic system disorders) | 6
lightheaded (Nervous system disorders) | 1
neutropenia (Blood and lymphatic system disorders) | 6
parotitis (Gastrointestinal disorders) | 1
proptosis (Eye disorders) | 1
sinus infection (Infections and infestations) | 1
strep throat (Infections and infestations) | 1
syncope (Nervous system disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 6
urinary tract infection (Infections and infestations) | 2
vasovagal (Nervous system disorders) | 1
weight gain (Investigations) | 1
wrist sprain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No